CLINICAL TRIAL: NCT05575986
Title: An Exploring Single Arm Study on the Efficacy and Safety of Herombopag Olamine in the Treatment of Thrombocytopenia After Chemotherapy in Malignant Tumors of the Digestive System
Brief Title: Herombopag Olamine in the Treatment of Thrombocytopenia After Chemotherapy
Acronym: hetrombopag
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xianglin Yuan, Chief physician, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR-OBU-HuB-CA-II-019
Record Dates: First submitted 2022-09-25; First posted 2022-10-12 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Malignant Tumors of the Digestive System; Trombocitopenia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Observation group (Experimental): Herombopag Olamine Tablets
  Interventions: Drug: Hetrombopag Olamine

INTERVENTIONS:
Drug: Hetrombopag Olamine — Hetrombopag Olamine 7.5mg orally, once a day, for 14 days. This product should be taken on an empty stomach, 2 hours after oral administration before eating, avoid taking it with meals.

SUMMARY:
To evaluate the efficacy and safety of hetrombopag in the treatment of thrombocytopenia after chemotherapy in patients with digestive system malignant tumors

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in clinical research and sign informed consent;
2. Age ≥18 years;
3. Digestive system malignancy confirmed by histology or cytology; Having used oxaliplatin combined with fluorouracil for at least one cycle of 21-day chemotherapy regimen (CAPOX or SOX regimen), platelet index after chemotherapy: ≥25×109/L and ≤75×109/L;
4. At least 10 days between TPO, IL-11 or platelet transfusion;
5. ECOG 0 to 2 points;
6. Expected survival time > 3 months;
7. Sufficient organ function for subsequent chemotherapy;
8. Women of reproductive age must be willing to use adequate contraception during the study of drug treatment.

Exclusion Criteria:

1. Thrombocytopenia caused by non-tumor chemotherapy drugs occurred within 6 months before screening, including but not limited to EDTA-dependent pseudothrombocytopenia, hypersplenism, infection, and bleeding;
2. Have any hematological malignancies, including leukemia, myeloma, bone marrow proliferative diseases, lymphoma or bone marrow proliferative diseases;
3. Clinically significant acute or active bleeding within the week prior to screening;
4. Subject has medically known hereditary prethrombotic syndrome (e.g., factor V Leiden mutation, prothrombin G20210A mutation, or hereditary antithrombin III (ATIII) deficiency)
5. The subject has a history of major cardiovascular disease (e.g., congestive heart failure (New York Heart Association Class 3/ cardiac function), known arrhythmias (e.g., atrial fibrillation) that increase the risk of thromboembolic events, coronary stenting, angioplasty, or coronary artery bypass grafting);
6. Subjects had a history of arterial or venous thrombosis within 3 months before screening;
7. Use of a vitamin K antagonist (including low molecular weight heparin, factor Xa inhibitor, or thrombin inhibitor) within 7 days prior to screening;
8. The subject has a history of chronic platelet or hemorrhagic disorders, or thrombocytopenia from causes other than CIT (e.g., chronic liver disease or immune thrombocytopenic purpura);
9. TPO, IL-11 or platelet infusion were used within 10 days before enrollment;
10. Previous use of thrombopoietin receptor agonists (e.g., eltrobopag, romiestine, etc.)
11. Those who cannot be treated with oral drugs;
12. Allergic to hetrombopag or any excipient;
13. Those whose organ function could not tolerate further antitumor therapy as assessed by the investigator; This product is not recommended for use or discontinuation of treatment in patients who meet any of the following criteria for liver function

ALT and AST > 8 x ULN.

ALT or AST>5×ULN for 2 weeks;

ALT or AST>3xULN (total bilirubin >2xULN or INR>1.5);

ALT or AST>3×ULN with progressive fatigue, nausea, vomiting, right upper abdominal pain or tenderness, fever, rash, and/or eosinophilia (>5%).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Days required for platelet recovery to ≥75×10^9/ L | At the end of Cycle 1 (each cycle is 28 days)
  Days required for platelet recovery to ≥75×10^9/ L

SECONDARY OUTCOMES:
The lowest platelet count | At the end of Cycle 2 (each cycle is 28 days)
  The lowest platelet count
Safety of treatment | 2 Cycle (each cycle is 28 days)
  Measure of time from study enrollment until progression.

CONTACTS AND LOCATIONS:
Locations (1):
- xianglin Yuan, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No